CLINICAL TRIAL: NCT05579275
Title: A Single-center, Open-label Study to Evaluate the Safety and Tolerability of JCXH-212 Monotherapy and Combined With Toripalimab in the Treatment of Malignant Solid Tumors
Brief Title: Evaluate the Safety and Tolerability of JCXH-212 Monotherapy and Combined With Toripalimab in the Treatment of Malignant Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, mingleizhuo, Chief Physician, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-JCXH-212-001
Record Dates: First submitted 2022-09-30; First posted 2022-10-13 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohort-experimental (Experimental): Patients will receive treatment for up to 1 year. Actual follow-up will be decided according to the patient 's condition and benefit, and each test requirement and data collection will be completed at specified time during the follow-up cycle.
  Interventions: Biological: JCXH-212 Injection

INTERVENTIONS:
Biological: JCXH-212 Injection — Based on the development principle of NCV, a community-type tumor neoantigen mRNA vaccine, JCXH-212 injection, has been developed that can be applied to patients with malignant solid tumors. NCVs activate tumor-specific CD4+ T cells and CD8+ T cells through active immunity, and these T cells can inhibit and kill tumor cells in cancer patients, thus prolonging the survival of cancer patients.

SUMMARY:
To evaluate the safety and tolerability of JCXH-212 monotherapy and combined with Toripalimab in patients with malignant solid tumors; to determine the maximum tolerated dose (MTD), and to evaluate the dose-limiting toxicity (DLT) of JCXH-212 monotherapy and combined with Toripalimab.

DETAILED DESCRIPTION:
This study uses 3+3 clinical design. About 12-24 patients with solid tumor malignancies are expected to be enrolled in this study.

For JCXH-212 monotherapy, 2 dose groups are set for dose escalation (100μg, 200μg). Doses were administered every 21 days, with a DLT observation period of 21 days after the first dose. After completion of DLT assessment, the investigator decided whether to continue the treatment after the end of DLT assessment based on the subject 's tolerance and the safety profile of the dose group. Subjects may continue to receive dosing if the investigator determines that the subject is benefiting from continued treatment. No more than 8 total doses of JCXH-212 will be administered.

For JCXH-212 combined with Toripalimab, 2 dose groups are set for dose escalation (100μg, 200μg of JCXH-212). JCXH-212 will be administered every 6 weeks, with a DLT observation period of 21 days after the first dose. Toripalimab (240mg per dose) will be administrated every 3 weeks. After completion of DLT assessment, the investigator decided whether to continue the treatment after the end of DLT assessment based on the subject 's tolerance and the safety profile of the dose group. Subjects may continue to receive JCXH-212 if the investigator determines that the subject is benefiting from continued treatment. No more than 8 total doses of JCXH-212 will be administered.

ELIGIBILITY:
Inclusion Criteria:

* The enrolled subjects shall meet all the following conditions at the same time:

  1. male or female patients, aged 18 ~ 75 years old;
  2. patients with advanced malignant solid tumors who have failed standard treatment (progression or intolerance after treatment) confirmed by pathology and/or cytology (only for Part 1);
  3. only for part2 : A. Patients with initial treatment, refusing or intolerant of standard treatment, PD-L1 (IHC 22C3) TPS ≥ 1%; B. Stage IIIB-IV patients with disease progression after previous standard treatment, who intend to receive immune monotherapy, can be enrolled regardless of the results of PD-L1; C. Stage II-III NSCLC patients after radical surgery, postoperative adjuvant chemotherapy (if necessary) has been completed, and PD-L1 (IHC 22c3) TPS is ≥ 1%, intend to receive adjuvant immunotherapy.
  4. tumor biopsy tissue samples can be provided for tumor neoantigen detection;
  5. ECOG (Eastern Cooperative Oncology Group) score of 0 ~ 1 in general condition;
  6. expected survival time of more than 3 months;
  7. patients have at least one measurable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECISTv1.1), the longest diameter at baseline is ≥ 10 mm (if lymph nodes, the short diameter is ≥ 15 mm);
  8. patients shall have sufficient bone marrow reserve function, and have no liver and kidney coagulation dysfunction, and laboratory test values shall meet the following conditions:

     1. absolute neutrophil count > 1.5 × 10/L, And white blood cell count > 3 × 10/L;
     2. platelet count > 80 × 10/L;
     3. hemoglobin > 90 g/L;
     4. serum creatinine < 1.5 × upper limit of normal (ULN) and creatinine clearance calculated by Cockroft-Gault formula > 30 mL/min;
     5. if there is no confirmed liver metastasis, AST, ALT < 2.5 × ULN; if there is confirmed liver metastasis, AST, ALT < 5 × ULN;
     6. if there is no liver metastasis, total bilirubin < 1.5 × ULN; if there is liver metastasis or Gilbert 's syndrome (hyperindirect bilirubinemia), total bilirubin < 3 × ULN;
     7. international normalized ratio (INR) < 1.5, and activated partial thromboplastin time (APTT) < 1.5 × ULN;
  9. tumor tissue gene detection suggests that one or more vaccines contain positive tumor neoantigen expression;
  10. patients do not have brain metastasis (except asymptomatic or stable brain metastasis after treatment for more than four weeks);
  11. Any adverse reactions caused by previous treatment must have recovered to grade 0-1 (except alopecia and vitiligo) within 4 weeks before the first dose of study drug;
  12. Patients voluntarily signed informed consent and expected compliance.

      Exclusion Criteria:
* Those meeting any of the following conditions may not be included.

  1. Known or suspected hypersensitivity to the ingredients of the study drug or its analogues;
  2. Only for Part 2: adverse reactions of grade ≥3 occurred after using ICIs in the past; except maculopapules /itching and reactive cutaneous capillary hyperplasia (RCCEP), there is no need to stop ICIs in hypothyroidism. Or those who are at high risk of receiving ICI treatment.
  3. Patients with any other disease or medical condition that is unstable or may affect their safety or study compliance, any serious or uncontrolled systemic disease, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, active gastrointestinal ulcers, abnormal immune function, etc.;
  4. Cardiovascular and cerebrovascular diseases/symptoms/indications that meet any of the following conditions:

     1. mean resting QTc > 470 ms (corrected QT interval [corrected by Fridericia formula]), mean QTc of 3 ECGs, QT interval measurement should start from QRS complex to the end of T wave);
     2. any clinically significant resting ECG abnormalities in rhythm, conduction or morphology, such as complete left bundle branch block, grade 2 and 3 heart block, PR interval > 250 ms, etc.;
     3. any factor that increases the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, etc. or unexplained sudden death in a first-degree relative under 40 years of age, or any concomitant medication known to prolong the QT interval;
     4. left ventricular ejection fraction (LVEF) < 50%;
     5. previous history of decreased myocardial contractility, i.e.Patients who presented with relevant symptoms within 6 months before study drug administration: such as chronic congestive heart failure, pulmonary edema or decreased cardiac ejection fraction;
     6. patients who had a history of acute or chronic cardiovascular and cerebrovascular diseases and presented with relevant symptoms within 6 months before study drug administration: myocardial infarction, severe or unstable angina pectoris, cerebral infarction, cerebral hemorrhage, or transient ischemic attack;
  5. . Patients who had an active second primary malignant tumor within 2 years before the first dose of study drug, except for specific cancers to be investigated and locally recurrent cancers that had undergone radical treatment (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ);
  6. . Patients with uncontrollable malignant third space effusion;
  7. . For women of childbearing age (postmenopausal women must have been postmenopausal for at least 12 months to be considered of non-childbearing potential), positive serum pregnancy test results within 7 days before the first dose of study drug;
  8. Have received major surgery within 4 weeks before the first administration of the study drug; Before receiving the study drug for the first time, the elution period for previous anti-cancer treatments (chemotherapy, targeted drugs, immunotherapy and radiotherapy) or any other study treatment is less than 3 weeks or 5 half-lives, whichever is shorter.
  9. Other serious, acute or chronic clinical or mental diseases or laboratory abnormalities that may increase the risk of research and drug use, or may interfere with the research results;
  10. patients with active autoimmune diseases or history of autoimmune diseases but may relapse, but patients with the following diseases are not excluded and can be further screened:

      1. type I diabetes;
      2. hypothyroidism (if controlled with hormone replacement therapy alone);
      3. controlled celiac disease;
      4. skin diseases that do not require systemic treatment (e.g., vitiligo, psoriasis, alopecia) ;
      5. any other disease that does not recur in the absence of external triggers;
  11. active human immunodeficiency virus (HIV), syphilis, hepatitis C virus (HCV) or hepatitis B virus (HBV) infection, asymptomatic chronic hepatitis B or C carriers can be excluded; active HBV, HCV and HIV infection is defined as:

      1. HBsAg positive and HBV DNA ≥ 1000 cps/ml (or 200 IU/ml);
      2. anti-HCV antibody and HCV RNA positive;
      3. HIV antibody positive;
  12. Active infection and need anti-infection treatment;
  13. Patients with a history of organ transplantation;
  14. Any form of primary immunodeficiency (such as severe combined immunodeficiency disease);
  15. Use of immunosuppressive drugs within 7 days before the first dose of study treatment, excluding: nasal spray, inhalation or other routes of local glucocorticoids or physiological doses of systemic glucocorticoids (that is, no more than 10mg/ day of prednisone or equivalent doses of other glucocorticoids); Short-term (≤7 days) use of prophylactic or therapeutic corticosteroids is allowed to avoid non-autoimmune allergic reactions (for example, pretreatment before intravenous contrast agent or drug administration);
  16. The investigator believes that the patient is not suitable for this trial for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity (DLT) | Up to 21 days after first dose every subject
  Tolerability and safety analysis: determine the maximum tolerated dose (MTD) and determine the escalation of the relevant dose. Incidence of DLTs was summarized overall and by dose level based on the DLT Analysis Set (DLTS).
analysis of primary efficacy indicators | At the end of the time 3-6 months after last subject last dose
  Efficacy analysis: In the study, correlation analysis will be performed between the main efficacy indicators and dose regimen in each dose group.

SECONDARY OUTCOMES:
exploratory analysis of changes in peripheral blood neoantigen-specific T cell responses before and after administration | The day of administration of the last subject
  Exploratory analysis: focus on describing changes in peripheral blood neoantigen-specific T cell responses before and after administration and the possible association or predictive role of such changes with treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo Minglei, Physician, Principal Investigator — Peking University Cancer Hospital & Institute; zhuo Minglei, Physician, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China